CLINICAL TRIAL: NCT02965547
Title: Remote Ischemic Preconditioning of Dynamic Cerebral Autoregulation in Healthy Adults
Acronym: RIPCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yi Yang (Other)
Responsible Party: Sponsor-Investigator, Yi Yang, Associated Dean of First Hospital of Jilin University, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RIPCA
Record Dates: First submitted 2016-11-14; First posted 2016-11-16 (Estimated); Last update posted 2021-08-24 (Actual); Status verified 2016-12

CONDITIONS: Ischemic Preconditioning
Keywords: Ischemic Preconditioning; dynamic cerebral autoregulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RIPC Group (Experimental): RIPC was induced by 4 cycles of extremities ischemia (5-minute blood-pressure cuff inflation to 200 mm Hg, followed by 5-minute cuff deflation).All subjects will take RIPC intervention, blood collection and 7 dCA measurements.
  Interventions: Device: Remote ischemic conditioning equipment; Procedure: Intravenous blood collection; Procedure: dCA measurement

INTERVENTIONS:
Device: Remote ischemic conditioning equipment — The RIPC consisted of 4 cycles of extremities ischemia (5-minute blood-pressure cuff inflation to 200 mm Hg, followed by 5-minute cuff deflation). The tourniquets were applied to one side upper arm and other side thigh. This intervention was undertaken one time in total.
Procedure: Intravenous blood collection — Nurses will collect intravenous blood 6ml twice(at baseline and 1h after RIPC).The blood samples will be stored for laboratory test.The blood samples only use for the trial.
Procedure: dCA measurement — Serial measurements of dCA were performed at 7 time points, baseline, 1h, 3h, 6h, 9h, 12h, 24h after RIPC.The continuous ABP was measured non-invasively using a servo-controlled plethysmograph (Finometer Pro, the Netherlands) at the middle finger. Two 2 MHz transcranial Doppler probe was used to measure continuous cerebral blood flow velocity (CBFV) simultaneously in the bilateral middle cerebral arteries at a depth of 45-60 mm Endtidal CO2 was monitored using a capnograph (MultiDop X2, DWL, Sipplingen, Germany). The probes were placed over temporal windows and fixed with a customized head frame. CBFV and continuous arterial blood pressure were recorded simultaneously from each subject in the supine position for 10 minutes. All data were recorded for further assessment and analysis.

SUMMARY:
The purpose of this study is to determine the impact of remote ischemic preconditioning on dynamic cerebral autoregulation and related hematology indexes in healthy adults.

DETAILED DESCRIPTION:
Remote ischemic preconditioning(RIPC) is the phenomenon whereby brief cycles of ischemia and reperfusion, applied to a distant organ, provide protection to the target organ. Dynamic cerebral autoregulation(dCA), a mechanism to maintain the cerebral blood flow, has been proved to be critical for the occurrence,development and prognosis of ischemic neurovascular disease. In this study, we hypothesis that RIPC provides neuro-protection by means of improving dCA.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 70,both genders
* Willing to participate in follow-up visits

Exclusion Criteria:

* current or having a history of chronic physical diseases or mental diseases
* suffering from infectious diseases in late one month
* pregnant and lactating women；
* smoking or drinking；
* inability to cooperate sufficiently to complete the dCA examination

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-07-25 (Actual)

PRIMARY OUTCOMES:
phase difference(PD) in degree | 2 days
  A dynamic cerebral auto-regulation parameter derived from transfer function analysis.Continuous cerebral blood flow velocities of bilateral middle cerebral artery will be assessed noninvasively using transcranial Doppler. Spontaneous arterial blood pressure will be simultaneously recorded using a servo-controlled plethysmograph on the left or right middle finger with an appropriate finger cuff size. Transfer function analysis will be used to derive the autoregulatory parameters.
the rate of recovery of cerebral blood flow velocity | 2 days
gain in cm/s/mmHg | 2 days

SECONDARY OUTCOMES:
resistance index (RI) changes from supine to upright position | 2 days
pulsatility index (PI) changes from supine to upright position | 2 days
mean middle cerebral artery blood flow velocity (mCBFV) changes from supine to upright position | 2 days

CONTACTS AND LOCATIONS:
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China

REFERENCES:
- [Derived] Qu Y, Liu J, Guo ZN, Zhang PD, Yan XL, Zhang P, Qi S, Yang Y. The Impact of Remote Ischaemic Conditioning on Beat-to-Beat Heart Rate Variability Circadian Rhythm in Healthy Adults. Heart Lung Circ. 2021 Apr;30(4):531-539. doi: 10.1016/j.hlc.2020.08.017. Epub 2020 Oct 5. PMID 33032892
- [Derived] Guo ZN, Guo WT, Liu J, Chang J, Ma H, Zhang P, Zhang FL, Han K, Hu HH, Jin H, Sun X, Simpson DM, Yang Y. Changes in cerebral autoregulation and blood biomarkers after remote ischemic preconditioning. Neurology. 2019 Jul 2;93(1):e8-e19. doi: 10.1212/WNL.0000000000007732. Epub 2019 May 29. PMID 31142636